CLINICAL TRIAL: NCT02430454
Title: Vignette-based Randomized Controlled Trial of the Decision Making Process of Bed Allocation in the Intensive Care Unit: Impact of Bed Availability and Cognitive Load.
Brief Title: Impact of Bed Availability and Cognitive Load on Intensive Care Unit Bed Allocation: a Vignette-based Clinical Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, João Gabriel Rosa Ramos, PhD Student, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 43084815.0.0000.0068
Record Dates: First submitted 2015-04-14; First posted 2015-04-30 (Estimated); Last update posted 2016-01-08 (Estimated); Status verified 2016-01

CONDITIONS: There Are no Specific Conditions Under Study; This Study Evaluates the Clinical Decision-Making Associated With Intensive Care Units Rationing
Keywords: ICU; decision making

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental (Experimental): Subjected to increased cognitive load
  Interventions: Behavioral: Increased cognitive load
- Control (No Intervention): Not subjected to increased cognitive load

INTERVENTIONS:
Behavioral: Increased cognitive load — simulated conditions to increase cognitive load: encourage first impression, time-limit, distractions
  Arms: Experimental

SUMMARY:
Decisions about ICU beds allocations are made everyday, specially in countries with scarcity of ICU beds, such as Brazil. ICU triage, most of the time, is not structured, which may lead to faulty decision making, possibly leading to bad clinical outcomes. It has been shown that external factors may influence the decision making process. The investigators intend to evaluate the impact of bed availability and cognitive load on the ICU bed allocation process by submitting groups of individuals to a vignette based randomized controlled trial simulating conditions with or without increased cognitive load and conditions with or without scarcity of ICU beds.

DETAILED DESCRIPTION:
Vignettes will be constructed based on consecutive patients for whom ICU bed was solicited. Vignettes will be validated through the evaluation of 8 experts in situations with or without bed scarcity. Vignettes with more than 80% concordance on ICU disposition (admission or refusion) will be used in the trial.

Intensive care doctors in Brazil will be asked to answer an online questionnaire with demographic characteristics and randomized to one of two groups. The experimental group will be submitted to increased cognitive load conditions, meaning that they will be encouraged to give their first impression on the vignettes, will have a time limit to answer the questions and will have popups with sound and videos, with the purpose to distract the respondents. The control group will be encouraged to think thoroughly and will have no time limit or distractions.

Vignettes will be presented, randomly, in conditions with or without scarcity of ICU beds to both groups. So, respondents with and without increased cognitive load will evaluate vignettes in conditions with and without scarcity of ICU beds.

ELIGIBILITY:
Inclusion Criteria:

* Intensive care unit doctors participating in specialty email lists

Exclusion Criteria:

* Consent not provided

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2015-04; Primary Completion 2015-11 (Actual); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
simulated ICU admission rates | 24 hours
  difference on simulated ICU admission rates between the experimental and control groups, comparing to the expected allocation (designated by the experts that validated the vignettes and Society of Critical Care Medicine priority rank)

SECONDARY OUTCOMES:
Time to complete the questionnaire | 60 minutes
  difference on time to complete the questionnaire between the two groups

CONTACTS AND LOCATIONS:
Overall Officials: Joao G Ramos, MD, Principal Investigator — Hospital das Clinicas da Faculdade de Medicina da Universidade de Sao Paulo